CLINICAL TRIAL: NCT01671241
Title: Heat Loss Prevention in Very Preterm Infants in Delivery Rooms: A Multicenter, Randomized, Controlled Trial of Polyethylene Occlusive Total Body Skin Wrapping
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Prevention
Other Study IDs: LossPreventionTotalBodyWrap
Record Dates: First submitted 2012-07-17; First posted 2012-08-23 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Hypothermia; Preterm Infant
MeSH Terms: conditions — Hypothermia; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Total body polyethylene wrap (body plus head) (Experimental): The entire body surface (body plus head) is covered by a polyethylene wrap
  Interventions: Device: Polyethylene wrap
- Polyethylene wrap (body) (Active Comparator): A polyethylene wrap covers the patient's body up to the neck
  Interventions: Device: Polyethylene wrap

INTERVENTIONS:
Device: Polyethylene wrap
  Arms: Total body polyethylene wrap (body plus head)
Device: Polyethylene wrap
  Arms: Polyethylene wrap (body)

SUMMARY:
Hypothermia after delivery is a world-wide problem associated with morbidity and mortality. The conventional approach of drying the baby with a pre-warmed towel and radiant warmers is unsuccessful in a large proportion of very preterm infants. Polyethylene occlusive skin wrapping covering the infant's body up to the neck will reduce postnatal heat loss in very preterm babies and represents the standard of care recommended by the International Guidelines for Neonatal Resuscitation. The use of a polyethylene head cap will also reduce heat loss 9 and its efficacy is comparable to that obtained with the wrap. However, the proportions of hypothermic infants at NICU admission (temperature <34°C) in the wrapped group (62%) as well as in the infants covered with a polyethylene cap (43%) remain high. The combination of body and head protection with a polyethylene wrap needs to be evaluated further. The investigators conducted a prospective, randomized, controlled trial in very preterm infants to evaluate whether a polyethylene total body wrapping (body plus head) prevents heat loss after delivery better than polyethylene occlusive wrapping.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants <29 weeks' gestation born in the study centers

Exclusion Criteria:

* Congenital anomalies with open lesions (e.g. gastroschisis, meningomyelocele) and babies whose delivery was not attended by the neonatal team

Ages: 1 Minute to 3 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2011-01

PRIMARY OUTCOMES:
Axillary temperature taken on admission to the NICU (immediately after total body wrap and wrap removal) and again 1 hour later

SECONDARY OUTCOMES:
Mortality prior to hospital discharge
Major brain injury
percentages of hyperthermic infants at NICU admission

CONTACTS AND LOCATIONS:
Locations (1):
- University of Padua, Azienda Ospedaliera di Padova, Padua, Italy

REFERENCES:
- [Background] Vohra S, Roberts RS, Zhang B, Janes M, Schmidt B. Heat Loss Prevention (HeLP) in the delivery room: A randomized controlled trial of polyethylene occlusive skin wrapping in very preterm infants. J Pediatr. 2004 Dec;145(6):750-3. doi: 10.1016/j.jpeds.2004.07.036. PMID 15580195
- [Background] Vohra S, Frent G, Campbell V, Abbott M, Whyte R. Effect of polyethylene occlusive skin wrapping on heat loss in very low birth weight infants at delivery: a randomized trial. J Pediatr. 1999 May;134(5):547-51. doi: 10.1016/s0022-3476(99)70238-6. PMID 10228287
- [Background] Trevisanuto D, Doglioni N, Cavallin F, Parotto M, Micaglio M, Zanardo V. Heat loss prevention in very preterm infants in delivery rooms: a prospective, randomized, controlled trial of polyethylene caps. J Pediatr. 2010 Jun;156(6):914-917.e1. doi: 10.1016/j.jpeds.2009.12.021. Epub 2010 Mar 15. PMID 20227728
- [Derived] Doglioni N, Cavallin F, Mardegan V, Palatron S, Filippone M, Vecchiato L, Bellettato M, Chiandetti L, Trevisanuto D. Total body polyethylene wraps for preventing hypothermia in preterm infants: a randomized trial. J Pediatr. 2014 Aug;165(2):261-266.e1. doi: 10.1016/j.jpeds.2014.04.010. Epub 2014 May 14. PMID 24837862